CLINICAL TRIAL: NCT03461471
Title: Exercise in All ChemoTherapy
Acronym: EnACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Kathryn Schmitz, Professor, Public Health Science, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00005664
Record Dates: First submitted 2017-07-25; First posted 2018-03-12 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Chemotherapy; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Exercise intervention
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Exercise intervention

SUMMARY:
Exercise in all Chemotherapy (EnACT) is a study to assess safety, feasibility, and acceptability of an exercise program within chemotherapy. This will be a single group study to capture the effects of an exercise intervention on the average chemotherapy patient and the patients compliance to the study.

DETAILED DESCRIPTION:
Several national and international agencies recommend exercise participation for all persons following a cancer diagnosis. The current evidence suggests that exercise training is safe during primary adjuvant therapy and improves physical function and quality of life outcomes. Moderate exercise has been shown to improve fatigue (extreme tiredness), anxiety, and self-esteem. It also helps heart and blood vessel fitness, muscle strength, and body composition. However, despite guidance on implementing exercise recommendations for cancer patients, exercise counseling is still not standard of care in cancer centers across the U.S. Our goal is to collect data that will assist with translation of the evidence from randomized clinical trials into standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥18 years of age
* Fluent in written and spoken English
* Must be able to provide and understand informed consent
* Must have an ECOG PS of ≤ 2
* Diagnosed with a solid tumor malignancy
* Cancer patients (stage 1-4)
* Scheduled to receive chemotherapy at Penn State Cancer Institute
* Absence of absolute contraindications for exercise according to the American Heart Association
* Primary attending oncologist approval

Exclusion Criteria:

* Receiving chemotherapy at a location other than Penn State Cancer Institute
* Not fluent in written and spoken English
* Hematological malignancy
* Evidence in the medical record of an absolute contraindication for exercise
* Cardiac exclusion criteria:

  * Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty or stenting within the past 6 months prior to the start of chemotherapy
  * Uncontrolled arrhythmias; patients with rate controlled atrial fibrillation for >1 month prior to start of chemotherapy may be eligible
  * syncope
  * acute myocarditis, pericarditis, or endocarditis
  * acute pulmonary embolus or pulmonary infarction
  * thrombosis of lower extremities
  * suspected dissecting aneurysm
  * pulmonary edema
  * respiratory failure
  * acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise
  * mental impairment leading to inability to cooperate
* Non-English speaking
* Pregnant women
* Children (the protocol will only include individuals 18 and older)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Assess Feasibility | Feasibility will be assessed at the completion of the study for each patient (average of 5 months of chemotherapy).
  Feasibility will be obtained if one third of chemotherapy patients actually do the exercise prescribed (one exercise session per week for four weeks).

SECONDARY OUTCOMES:
Compare changes in pain, physical function, nausea, vomiting, arthralgias, chemotherapy alterations (dose delays and alterations). | Surveys will be given once the patient is consented and again at the completion of the study for each patient (average of 5 months per patient).
  This will be compared using surveys at the beginning and end of chemotherapy (or intervention). Data will also be collected on the initial chemotherapy prescription and whether there are dose alterations.
Qualitative assessments of clinician perspectives regarding the study. At the end of the study clinicians will be asked a series of qualitative questions to gain their insight into the study. | Surveys will be provided to clinicians at the completion of the study (up to 38 months)
  At the conclusion of the study, clinicians within the institution will be asked qualitative questions regarding the study.
Assessing safety through number of patients with injuries related to the intervention | A standardized survey for assessing injuries will be used and administered at the end of the patients chemotherapy (average of 5 months)..
  The investigator will be using a standardized Adverse Events/Injury History survey as the primary instrument in assessing safety. This survey focuses on asking questions to gauge the participants experience with muscle strain, joint pain, among other things, in order to assess if there were any complications associated with the intervention. The investigator will consider the intervention safe if less than 25% of included patients report mild musculoskeletal impairments and less than 5% experienced musculoskeletal injuries (defined as symptoms lasting a week or longer and or requiring the attention of a medical professional).
Assess Acceptability | Acceptability will be assessed at the completion of the study for each patient (average of 5 months of chemotherapy).
  We will consider the intervention to be acceptable if more than 50% of the patients approached agree to receive at least the first session of exercise counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Cancer Institute, Hershey, Pennsylvania, United States